CLINICAL TRIAL: NCT04778371
Title: The Effects of Almond Consumption on Functional Performance, Aerobic Capacity, and Physical Activity in Overweight Active Older Adults
Brief Title: The Effects of Almond Consumption on Functional Performance and Activity in Overweight Active Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Bob Hickner, Principal Investigator, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 00001394
Record Dates: First submitted 2021-01-27; First posted 2021-03-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Overweight
Keywords: almond; functional performance; aerobic capacity; physical activity
MeSH Terms: conditions — Overweight; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, calorie-match controlled, crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond supplement (Experimental): Participants will consume 32 g dry roasted, unsalted almonds twice a day for 12 weeks
  Interventions: Other: Almonds
- Placebo matched supplement (Placebo Comparator): Participants will consume 100 g granola bar, calorie matched to Almond, twice a day for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Almonds — 64 g total dry roasted, unsalted almonds per day for a total of 12 weeks
  Arms: Almond supplement
Other: Placebo — 200 g total calorie matched granola bar per day for total of 12 weeks
  Arms: Placebo matched supplement

SUMMARY:
The overall objective of this proposed randomized, crossover study is to determine the effect of 12 weeks of almond consumption, ingested as a snack twice daily, on energy expenditure, performance and functional related outcomes, in active, overweight, older adults, in comparison to 12 weeks of an isocaloric matched control snack. The central hypothesis of this study is, due to the nutritionally beneficial composition of almonds, that daily consumption of an almond snack for 12 weeks will contribute to improvements in energy expenditure, physical and functional performance, vascular function, inflammation/oxidative stress, sleep quality, mood status, and body composition in active, overweight and obese older adults compared to an isocaloric commercially available snack.

DETAILED DESCRIPTION:
By 2030 it estimated that 20% of individuals in the United States (U.S.) will be 65 years of age or older, indicating a shift in demographics over the past century. The aging process is strongly associated with reduced aerobic capacity and functional performance as well as increases in inflammation and oxidative stress. With differences in the demographic profile, eating patterns have also changed for Americans within the past 30 years, with a majority of Americans consuming at least one snack/day; with the types of snacks consumed being processed foods that are high in refined carbohydrates, saturated fats, and low in fiber. Additionally, the aging process contributes to decreases in RMR, which can promote alterations in body composition. Lifestyle modifications have been shown to contribute to beneficial outcomes associated with aging. Therefore, healthy, nutrient-dense foods are of primary importance for enhancing functional performance, aerobic capacity, and physical activity as well as improving vascular function, body composition, and markers of inflammation/oxidative stress within this growing population. Tree nuts are a nutrient- and energy dense food, which may contribute to increases in RMR due to their high amounts of poly- and monounsaturated fatty acids affecting diet-induced thermogenesis. Almonds (Prunus dulcis) are an excellent source of α-tocopherol and a good source of monounsaturated fat, magnesium, fiber, and protein. When compared to other nuts almonds have the greatest amount of fiber and protein. Almond supplementation has been shown to attenuate age-related decline in aerobic fitness and physical performance measures. Few studies have assessed how almonds alone affect fitness and physical function. However, Yi et al. found that in young healthy, endurance trained individuals, consumption of almonds elevated serum arginine, nitric oxide and TAC, all of which contributed to improved exercise performance. Constituents of almonds including L-arginine and magnesium have been shown to increase anaerobic threshold and physical performance in healthy active older adults respectively . Studies have found that the incorporation of almonds in a diet can decrease oxidative stress and improve vascular function. Improvements in both FMD and systolic blood pressure were shown after 4 weeks of almond consumption in healthy old and young men. L-arginine, an amino acid vital for synthesis of nitric oxide, which controls vascular tone, is also found in almonds. Almonds are often cited as a healthy, protein-boosting snack, beneficial for sustaining muscle mass and metabolism, without increasing fat mass or total energy intake. Additionally, studies have demonstrated that body weight and body mass index (BMI) remain unchanged during almond supplementation interventions. Almond consumption has also been shown to decrease visceral fat and body fat percentage. The extent to which daily almond consumption affects functional performance, aerobic capacity, energy expenditure, vascular function, body composition and inflammation/oxidative stress in active overweight and obese older adults needs to be investigated.

For this study, fifty men and postmenopausal women will follow a randomized-controlled crossover design. If individuals qualify for participation after the screening visit, they will be asked to complete a 3-day food record and wear an ActiGraph to track physical activity and sleeping patterns for the next seven days, to be returned at their Baseline Study Visit #1. During the Baseline Study Visit #1 assessments of: RMR, body composition (DXA), vascular assessments (FMD, PWV, PWA, blood pressure), heart rate, anthropometrics (height, weight, and waist/hip circumference), venous blood draw, POMS, and sleep quality (PSQI) will be collected. The following day, participants will return for their Baseline Physical Performance Visit #1 to complete assessments of submaximal aerobic capacity and the CS-PFP. Following this visit, participants will be provided with 12 weeks of almonds or the isocaloric snack. Participants will be asked to come in after 6 weeks to receive the rest of their dietary regimen and to monitor compliance. During week 11, participants will be asked to come to the study site to be given a 3-day food record and the ActiGraph to be retuned at the Post-Test Study Visit #1. After 12 weeks, participants will return to FSU to complete their Post-Test Study Visit #1, which will involve all the same assessments from the baseline study visit, as well as their Post-Test Physical Performance Visit #1, the next day. After the 4-week washout period, participants will similarly be asked to complete a 3-day food record and wear an ActiGraph for the following 7 days, to be returned upon the participants' Baseline Study Visit #2, where participants will crossover into receiving the corresponding dietary regimen and will follow the same procedures for the following 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 50 physically active men and postmenopausal women (free of menstruation for 12 consecutive months)
* Between the ages of 50-59 years
* Free of any chronic diseases such as cancer
* Active lifestyle (>30 minutes, 3 days/week)
* BMI of 25.0 kg/m2 to 29.9 kg/m2 will be included
* There will be no restrictions based on race, ethnicity, or socioeconomic status.

Exclusion Criteria:

* Individuals diagnosed with cardiovascular diseases (CVD) Type 2-diabetes
* Uncontrolled hypertension (≥160/100 mmHg)
* BMI <25.0 kg/m2 or >29.9 kg/m2
* Other active chronic diseases such as cancer, asthma, glaucoma, kidney, liver and pancreatic disease
* Those who are not post-menopausal or on hormone replacement therapy
* Taking more than one anti-hypertensive or have been taking them for less than 3 months -Any musculoskeletal or orthopedic problem that would otherwise prevent completing the study Participants participating in a weight loss program or having lost or gain ≥10% bodyweight within the last 6 months
* Currently using tobacco
* Consumption of >12 alcoholic drinks/week
* Nut allergies
* Frequent tree nut consumers (>2 servings/week)
* In concurrent participation with another investigational study
* Currently consuming any performance supplement (i.e. creatine, nitric oxide, whey/casein protein, branched chain amino acids).

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Effect of almonds on functional performance | 1 year
  Functional performance assessed by the Continuous-Scale Physical Functional Performance Test.
Effect of almonds on submaximal aerobic capacity (VO2) | 1 year
  -treadmill test ending at 85 % max VO2 measured using ParvoMedics metabolic cart with VO2 units reported in ml/(kg*min)-1

SECONDARY OUTCOMES:
Effect of almond on resting metabolic rate (RMR) | 1 year
  Resting metabolic rate as measured using the Parvomedics Metabolic Cart with resting metabolic rate being reported as VO2 in liters/minute.
Effect of almond on body fat | 1 year
  measured by duel energy x-ray absorptiometry and body fat reported as a percentage of total mass, in units of %.
  -
Effect of almond on lean body mass | 1 year
  measured by duel energy x-ray absorptiometry and reported as lean body mass in kilograms.
Effect of Almond on sleep pattern | 1 year
  Actigraph watch worn for 1 week prior to baseline and post-tests
  -monitors sleep activity and reported in units of minutes.
Effect of Almond on arterial health using flow mediated dilation | 1 year
  Measure of flow-mediated dilation (FMD) via use of the Philips HD11XE Doppler Ultrasound, which measures the ability of an artery to expand (dilate) in response to sheer stress caused by an increase in blood flow.
  -Brachial artery FMD will be examined using a linear array transducer and will be reported in units of %.
Effect of Almond on arterial health using pulse wave velocity | 1 year
  -Measured using the Automated Pulse-Wave Velocity (PWV) Device (VP-2000, Omron Healthcare Inc.) with PWV being the velocity at which the blood pressure pulse is conducted through the circulatory system via an artery or a combined series and length of arteries. Used to measure arterial stiffness and reported in units of m/sec.
C-reactive protein | 1 year
  Measured via fasting blood draw 20 ml using ELISA analyses and reported in units of nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hickner, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States